CLINICAL TRIAL: NCT05249218
Title: Impact of Fruits and Vegetables on Metabolic Control in Children With PKU
Brief Title: Impact of Fruit and Vegetables in PKU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alex Pinto (Other)
Responsible Party: Sponsor-Investigator, Alex Pinto, Research Dietitian, Birmingham Children's Hospital, United Kingdom
Organization: Birmingham Children's Hospital, United Kingdom (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 18/BC/DTS/NO/215
Record Dates: First submitted 2021-06-10; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Phenylketonurias
Keywords: Fruit and vegetables; Phenylalanine; Animal protein; Vegetable protein
MeSH Terms: conditions — Phenylketonurias | interventions — Yogurt

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomised controlled study over 21 weeks in children to assess how Phe intake from fruits and vegetables (containing 76-100 mg Phe/100g) vs. animal sources will impact on blood Phe control. This will be followed by a 6 months extension study examining the 'unlimited' use of fruits and vegetables containing Phe 76-100 mg/100g on blood Phe control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group starting intervention with vegetable protein (Active Comparator): Phase A followed by Phases B, C, D, E.
  Interventions: Other: Phase B - Extra 1 Phe exchange from fruits/vegetables containing Phe from 76-100mg/100g; Other: Phase C - Extra 2 Phe exchanges from fruits/vegetables containing Phe from 76-100mg/100g; Other: Phase D - Extra 1 Phe exchange from milk or yoghurt; Other: Phase E - Extra 2 Phe exchanges from milk or yoghurt
- Group starting intervention with animal protein (Active Comparator): Phase A followed by Phases D, E, B, C.
  Interventions: Other: Phase B - Extra 1 Phe exchange from fruits/vegetables containing Phe from 76-100mg/100g; Other: Phase C - Extra 2 Phe exchanges from fruits/vegetables containing Phe from 76-100mg/100g; Other: Phase D - Extra 1 Phe exchange from milk or yoghurt; Other: Phase E - Extra 2 Phe exchanges from milk or yoghurt

INTERVENTIONS:
Other: Phase B - Extra 1 Phe exchange from fruits/vegetables containing Phe from 76-100mg/100g — Usual low Phe diet + 60g fruits/vegetables containing Phe from 76-100mg/100g
Other: Phase C - Extra 2 Phe exchanges from fruits/vegetables containing Phe from 76-100mg/100g — Usual low Phe diet + 120g fruits/vegetables containing Phe from 76-100mg/100g
Other: Phase D - Extra 1 Phe exchange from milk or yoghurt — Usual low Phe diet but 1 x 50 mg extra Phe exchange from milk or yoghurt
Other: Phase E - Extra 2 Phe exchanges from milk or yoghurt — Usual low Phe diet but 2 x 50 mg extra Phe exchange from milk or yoghurt eaten daily

SUMMARY:
In the UK, some fruits and vegetables are permitted without measurement in the diets of people with phenylketonuria (PKU). It is proven that fruits and vegetables containing phenylalanine (Phe) up to 75mg/100g (e.g. carrots, sweet potato, tomatoes) do not affect blood Phe control but it is unknown to what extent fruits and vegetables containing Phe from 76-100mg/100g (e.g. cauliflower, broccoli, beansprouts and asparagus) increase blood Phe levels. In addition, there is very little information about how differently animal and vegetable protein affect blood Phe levels. It is believed that plant protein may have less bioavailability and therefore have less impact on blood Phe control. The investigators aim is to perform a randomized controlled study over 21 weeks in children (5-12y) with PKU. Children will be studied during five different time periods, examining the effect on blood Phe control when increasing Phe intake from vegetables/fruits containing Phe from 76-100 mg/100g vs. animal sources. At the end of the study, fruits and vegetables containing 76- 100mg Phe/100g will continue to be given as "exchange-free" for 6 months. This is a practical, cost effective study and should bring benefit to all people with PKU following a very restrictive diet both within the UK and throughout the world.

ELIGIBILITY:
Inclusion Criteria:

* PKU patients diagnosed by NBS and BH4 deficiencies;
* Early and continuously treated;
* Adherent to their prescribed PKU diet consisting of a protein-restricted diet and Phe-free amino acid based protein substitute;
* In good general health as evidenced by medical history;
* Able to provide written informed consent/assent (parent/child);
* Able to comply with the study protocol and take study product according to the opinion of the PI;
* Patients with good metabolic control (age 5-12y, 120-360μmol/L) with 3 out of 4 levels within range prior to consent (if 2 of 4 above target range but one close to the upper limit, PI to decide if patient can enter the study).

Exclusion Criteria:

* Concomitant diseases / disorders such as renal or gut disease / disorders and diabetes;
* Dislikes fruits and vegetables containing 76-100 mg of Phe/100g e.g.brocolli or cauliflower;
* Treated with BH4 (sapropterin);
* Presence of intercurrent infection;
* Patients with poor metabolic control (age 5-12y, >360μmol/L).

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Blood Phe levels three times a week of patients with PKU taking extra 1 or 2 exchanges of fruits and vegetables containing 76-100mg of Phe/100g during 4 weeks each. | 8 weeks
Blood Phe levels three times a week of patients with PKU taking extra 1 or 2 exchanges of animal protein during 4 weeks each. | 8 weeks

SECONDARY OUTCOMES:
Blood Phe levels three times a week with PKU taking fruits and vegetables containing 76-100mg of Phe/100g without measurement during 6 months. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Birmingham Women's and Children's Hospital, Birmingham, West Midlands, United Kingdom